CLINICAL TRIAL: NCT06689475
Title: The Effect of Simulation on Cardiac Auscultation Competence of Nursing Students: A Randomised Controlled Study
Brief Title: The Effect of Simulation on Cardiac Auscultation Competence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Evrim Eyikara, PhD, Gazi University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: GaziU-HF-ES-02
Record Dates: First submitted 2024-11-13; First posted 2024-11-14 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Auscultation of Heart; Simulation Based Learning; Psychoacoustics
Keywords: auscultation of cardiac sounds; Simulation; psychoacoustic; nursing students

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Psychoacoustic group (Experimental): The psychoacoustic approach group will listen to normal heart sounds (S1, S2), abnormal heart sounds (S3, S4) and murmur sounds from the audio file uploaded to their mobile phones in the laboratory environment through headphones for 500 repetitions each.
  Interventions: Other: Psychoacoustic approach
- Simulation group (Experimental): The simulation group will practice auscultation of heart sounds in a one-to-one and repetitive manner, working with a high reality simulator. Trainers will act as facilitators during the cardiac auscultation practice of the students in the intervention groups.
  Interventions: Other: Simulation
- Control group (No Intervention): The control group will continue with the standard education.

INTERVENTIONS:
Other: Psychoacoustic approach — The psychoacoustic approach group will listen to normal heart sounds (S1, S2), abnormal heart sounds (S3, S4) and murmur sounds from the audio file uploaded to their mobile phones in the laboratory environment through headphones for 500 repetitions each.
  Arms: Psychoacoustic group
Other: Simulation — The simulation group will practice auscultation of heart sounds in a one-to-one and repetitive manner, working with a high reality simulator. Trainers will act as facilitators during the cardiac auscultation practice of the students in the intervention groups.
  Arms: Simulation group

SUMMARY:
This randomized controlled study aims to determine the effect of simulation on the cardiac auscultation competence of nursing students. The main questions it aims to answer are:

* Simulation is effective in developing the cardiac auscultation competence of nursing students.
* The psychoacoustic approach is effective in developing the cardiac auscultation competence of nursing students.

One week after the 2-hour theoretical lecture, all three groups will be taken simultaneously to a 3-hour laboratory practice for cardiac auscultation. An instructor will lead each group to ensure coordination. The psychoacoustic approach group will listen to normal heart sounds (S1, S2), abnormal heart sounds (S3, S4) and murmur sounds from the audio file uploaded to their mobile phones in the laboratory environment through headphones for 500 repetitions each. The simulation group will practice auscultation of heart sounds in a one-to-one and repetitive manner, working with a high reality simulator. Trainers will act as facilitators during the cardiac auscultation practice of the students in the intervention groups. The control group will continue with the standard education.

ELIGIBILITY:
Inclusion Criteria:

- First-time registration in the course.

Exclusion Criteria:

* Non-native speakers of the country's native language.
* Previous graduation from any health-related university.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2024-12-25 (Actual); Primary Completion 2025-05-05 (Actual); Study Completion 2025-05-20 (Actual)

PRIMARY OUTCOMES:
achievement test | From enrollment to the end of education at 4 weeks.
  It is a four-question test in which students mark the cardiac sounds they listen to on the computer.

SECONDARY OUTCOMES:
Student Satisfaction and Confidence in Learning | At the end of education at 4 weeks.
  It is a five-point Likert-type scale consisting of 13 statements. It consists of two sub-dimensions: 'satisfaction with learning' and 'self-confidence'. The higher mean score obtained from the scale, the higher the student's satisfaction with the teaching method applied and the higher the level of self-confidence in learning.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University Faculty of Nursing, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No